CLINICAL TRIAL: NCT06921499
Title: Continuing and Expanding Va Meh Du, A Mental Health Promotion Program for Karenni Refugee Children and Emerging Adults
Brief Title: Va Meh Du: A Sports-based Mental Health Promotion Intervention for Karenni Refugees
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Greensboro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: UNCGreensboro
Record Dates: First submitted 2025-04-02; First posted 2025-04-10 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Coping Skills; Social Connectedness; Psychological Well Being; Physical Activity
Keywords: mental health education; sports-based mental health; mental health intervention; refugee health
MeSH Terms: conditions — Psychological Well-Being; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mental Health Education (Experimental)
  Interventions: Behavioral: Va Meh Du (Mental Health Education)
- Comparison (Active Comparator): Participants randomized to comparison will receive 20-30 minutes of team-building activities each week for roughly 5 weeks.
  Interventions: Behavioral: Active Compartor

INTERVENTIONS:
Behavioral: Va Meh Du (Mental Health Education) — Participants randomized to Va Meh Du (mental health education) will receive 20-30 minutes of mental health education each week for roughly 5 weeks. Mental health education will be evidence-based, using sports psychology practices, and culturally targeted toward Karenni refugees.
  Arms: Mental Health Education
Behavioral: Active Compartor — Participants randomized to comparison will receive 20-30 minutes of team-building activities each week for roughly 5 weeks.
  Arms: Comparison

SUMMARY:
The goal of this clinical trial is to learn if a soccer program focused on mental health positively impacts mental health in Karenni refugee young boys and men. The main questions it aims to answer are:

Does mental health education provided during a sports program improve mental health coping for Karenni refugee young boys and men? Does participation in a sports-program improve social connection for Karenni refugee young boys and men?

Researchers will compare those receiving mental health education to a comparison group to see if mental health education improves mental health coping skills.

Participants will:

Participate weekly soccer practices for 6 months Receive mental health education or comparison activities Answer questions about their health, such as their coping skills, social connection, and physical activity

ELIGIBILITY:
Inclusion Criteria:

* For child/minor participants: 8-16 years old, self-identifies as Karenni, self-identifies as a boy, speaks English, currently lives in Piedmont Triad area of NC, has parental consent, assents to participate
* For adult participants--18 years of age, self-identifies as Karenni, self-identifies as a man, speaks English and Karenni, currently lives in Piedmont Triad area of NC, consents to participate, anticipates missing no more than 2 practices

Exclusion Criteria:

* [for adult participants only]: Criminal record indicating potential harm to children (i.e., convicted of a violent or sexual crime, registration in the Sex Offender Registry, Responsible Individual List, or Child Maltreatment Registry) or are expected to miss more than 2 practices

Min Age: 8 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-17 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Coping Skills | From enrollment to end of intervention at 6 months
  Change in engagement coping skills will be measured using Coping Strategies Inventory-Short Form for adult participants and KIDCOPE for minor participants
Social Connectedness | From enrollment to end of intervention at 6 months
  Change in social connectedness will be measured using Social Connectedness Revised Scale for adult participants and NIH Toolbox Pediatric social relationship scales (Friendship and Loneliness) for minor participants

SECONDARY OUTCOMES:
Psychological Well being | From enrollment to end of intervention at 6 months
  Change in psychological well-being will be measured using the Flourishing Scale and WHO-5 for adult and minor participants
Physical Activity | From enrollment to end of intervention at 6 months
  Change in physical activity will be measured via the self-report questions: "In the past 3 months, how physically active have you been?" and "In the past 6 months, how physically active have you been?" Participants will answer using a 5-point Likert Scale from 1 (Very often) to 5 (Never).

CONTACTS AND LOCATIONS:
Locations (1):
- Bamboo Roots, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 12 months
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in IRB-approved research and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact adsucaldito@uncg.edu